CLINICAL TRIAL: NCT06175273
Title: The Pediatric Oncology Interventional Nutrition Therapy (POINT) Trial: A Pilot Study
Brief Title: Pediatric Oncology Nutrition Intervention Trial
Acronym: POINT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Corey Hawes (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Corey Hawes, Clinical Nutrition Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 89377; UL1TR001998 (NIH)
Record Dates: First submitted 2023-11-21; First posted 2023-12-18 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Cancer; Nutrition Related Cancer; Nutrition Aspect of Cancer; Muscle Loss; Malnutrition, Child
MeSH Terms: conditions — Neoplasms; Muscular Atrophy; Child Nutrition Disorders | interventions — Enteral Nutrition; Cyproheptadine; Olanzapine; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control (Active Comparator): Standard of Care who have either weight gain, weight maintenance, or weight loss <10%.
  Interventions: Other: Standard of Care
- Oral Nutrition Supplements (Experimental): Those receiving ONS will be prescribed a standard ONS (1.0 kcal per mL) that will meet a minimum of 50% of estimated energy needs to promote weight gain but allow for continued regular dietary intakes. The ONS will be prescribed as 8oz (240mL) per dose at least once a day, but up to six times per day depending on estimated nutrient needs.
  Interventions: Dietary Supplement: Oral Nutrition Supplement
- Enteral Nutrition (Experimental): Those randomized to EN will have a feeding tube placed and started on tube feeds via a designated pump for overnight feeds, meeting at least 50% of estimated energy needs to allow for continued regular dietary intakes during the day.
  Interventions: Dietary Supplement: Tube Feed
- Appetite Stimulants (Experimental): Those receiving age-appropriate appetite stimulants will be provided either cyproheptadine or olanzapine. Subjects will be given cyproheptadine if they fall between the ages of 2-12 years of age and olanzapine if they are >12 years of age or older.
  Interventions: Drug: Cyproheptadine; Drug: Olanzapine

INTERVENTIONS:
Dietary Supplement: Oral Nutrition Supplement — 8oz (240mL) per dose at least once a day, but up to six times per day depending on estimated nutrient needs. The formula will equate to 1.0kcal/mL
  Arms: Oral Nutrition Supplements
Dietary Supplement: Tube Feed — EN will have a feeding tube placed and started on tube feeds via a designated pump for overnight feeds, meeting at least 50% of estimated energy needs
  Arms: Enteral Nutrition
Drug: Cyproheptadine — 0.25mg/kg/d divided BID. May titrate by 4mg increments to a max of 12mg/day.
  Arms: Appetite Stimulants
Drug: Olanzapine — 2.5mg once a day (at night). May titrate by 2.5mg increments to max of 10mg/day
  Arms: Appetite Stimulants
Other: Standard of Care — Diet education on high protein, high calorie food consumption
  Arms: Control

SUMMARY:
Nearly 60% of pediatric patients diagnosed with cancer develop malnutrition caused by a combination of disease burden, side effects of chemotherapy, and the intensity of cancer treatment. These patients are known to have an increased risk of infection, treatment-related toxicity, inferior clinical outcomes, and increased risk of mortality. Malnutrition may progress to cancer cachexia, characterized by anorexia, increased inflammation, decreased fat, and decreased muscle mass with subsequent weight loss, which is associated with decreased overall survival.

The goal of the proposed research is to determine changes in body composition, weight status, and nutritional status between common nutrition interventions including oral nutrition supplements (ONS), appetite stimulants, and enteral nutrition (EN) among pediatric cancer patients. A secondary goal of this research is to utilize the findings to develop clinical nutrition guidelines for this patient population. The specific objective of the research proposed is to solve the lack of evidence to adequately treat nutritional deficits in the pediatric oncology population. Without this data, there is a lack of clinical consistency in the initiation and selection of appropriate nutrition interventions to provide a more definitive pathway of care. This study can help formulate a clinical guideline for this patient population before, during, and after treatment.

DETAILED DESCRIPTION:
The investigators plan to enroll a minimum of 45 subjects between the ages of 2-18 years old, over the course of one year, including males and females of all ethnicities. The subject will be a newly diagnosed pediatric patient with cancer who will actively receive chemotherapy at UK Healthcare's Kentucky Children's Hospital (KCH).

All those who enroll will have a baseline ultrasound and biomarkers taken at enrollment. Participants will also receive 'standard of care' medical nutrition therapy (MNT) counseling at diagnosis for following a high protein/high-calorie diet. If any of the enrolled participants lose >10% of the diagnosis weight, the participants will then be randomized to receive (1) oral nutrition supplements, (2) age-appropriate appetite stimulants, or (3) enteral nutrition via a feeding tube. At the point of randomization, participants will receive another ultrasound and biomarkers. Those randomized will then receive additional ultrasounds and biomarkers at 1 month and 3 months after randomization. The remaining patients that have either weight maintenance or weight gain, will be utilized as a comparator group and will receive an ultrasound at 3 months and 6 months from enrollment/diagnosis. Each group will have a goal of at least 10 patients per group.

Those receiving ONS will be prescribed a standard ONS (1.0 kcal per mL) that will meet a minimum of 50% of estimated energy needs to promote weight gain but allow for continued regular dietary intakes. The ONS will be prescribed as 8oz (240mL) per dose at least once a day, but up to six times per day depending on estimated nutrient needs. Those receiving age-appropriate appetite stimulants will be provided either cyproheptadine or olanzapine. Subjects will be given cyproheptadine if the participants fall between the ages of 2-12 years of age and olanzapine if the participants are >12 years of age or older. Table 1 summarizes the medication dosage forms, initial and dose titration options, and precautions/contraindications of each appetite stimulant. Medication adjustments will be made within 2-4 weeks of initiation due to the variable peak effect times, and chemotherapy treatment plans dictating clinic follow-up. Those randomized to EN will have a feeding tube placed and started on tube feeds via a designated pump for overnight feeds, meeting at least 50% of estimated energy needs to allow for continued regular dietary intakes during the day. After placement of a feeding tube, an abdominal x-ray will be obtained per hospital policy to confirm the appropriate placement of the feeding tube prior to use to ensure the safety of using said feeding tube.

Baseline demographics will be collected, including gender, age, diagnosis, QMLT ultrasound measurement, subjective global assessment (SGA) malnutrition risk, pediatric z-scores, and activity levels. Investigators will assess the subjects' nutritional intake, body composition via QMLT ultrasound, mid-upper arm circumference, pediatric z-scores (weight, length, and body mass index), biomarkers (leptin, IL-6, Lipid profiles, Cystatin-C, Vitamin D, and C-reactive protein), compliance and tolerance to nutrition intervention, physical activity, and clinical outcomes (rates of infection, number of hospital days for non-chemotherapy administration, number of clinic visits for non-chemotherapy administration, chemotherapy toxicity CTCAE grade, rate or relapse, and 1-year survival rates) at multiple time points throughout the study. Nutritional assessment will involve a 24-hour food recall which will be performed at diagnosis, randomization, and then every 1-2 weeks once randomized to an intervention. Weight loss and pediatric z-scores (weight-for-age, length-for-age, and BMI-for-age) will be assessed every 1-2 weeks throughout the study enrollment. Ultrasound assessment will be of the QMLT by measuring at the midpoint between the ASIS and the upper pole of the patella. The measurements will be taken bilaterally, three times, and averaged together for the final measurement. Ultrasound assessment will occur at enrollment when weight loss criteria are met for randomization, and then at 1 month and 3 months after randomization (or when the weight lost is regained).

Pediatric physical activity will be assessed every 1-2 weeks in combination with ultrasound measurements. Adherence and adverse effects to medications, tube feeds, or oral nutrition supplements will be assessed at each clinic visit. Biomarkers will be analyzed at randomization, 1 month, and 3 months after randomization.

Standard of care for patients are to receive MNT education at diagnosis. For those that lose weight, standard of care is to receive the nutrition interventions listed above (oral nutrition supplements, appetite stimulants, or enteral nutrition via feeding tube). The standard of care is to generally go from a least invasive to a more invasive approach. The research components of this study include being randomized to a nutrition intervention rather than a non-validated step-wise approach, the ultrasound measurements, and the biomarkers. These components are not considered standard of care and are research procedures. Baseline demographics will be collected, including gender, age, diagnosis, QMLT ultrasound measurement, subjective global assessment (SGA) malnutrition risk, pediatric z-scores, and activity levels. The team will assess the subjects' nutritional intake, body composition via QMLT ultrasound, mid-upper arm circumference, pediatric z-scores (weight, length, and body mass index), biomarkers (leptin, IL-6, Lipid profiles, Cystatin-C, Vitamin D, and C-reactive protein), compliance and tolerance to nutrition intervention, physical activity, and clinical outcomes (rates of infection, number of hospital days for non-chemotherapy administration, number of clinic visits for non-chemotherapy administration, chemotherapy toxicity CTCAE grade, rate or relapse, and 1-year survival rates) at multiple timepoints throughout the study. Nutritional assessment will involve a 24-hour food recall which will be performed at diagnosis, randomization, and then every 1-2 weeks once randomized to an intervention. Weight loss and pediatric z-scores (weight-for-age, length-for-age, and BMI-for-age) will be assessed every 1-2 weeks throughout the study enrollment. Ultrasound assessment will be of the QMLT by measuring at the midpoint between the ASIS and the upper pole of the patella, a total of 4 ultrasounds will be conducted during the study. The measurements will be taken bilaterally, three times, and averaged together for the final measurement. Ultrasound assessment will occur at enrollment when weight loss criteria are met for randomization, and then every 1-2 weeks for up to 8 weeks after randomization. Pediatric physical activity will be assessed every 1-2 weeks in combination with ultrasound measurements. Adherence and adverse effects to medications, tube feeds, or oral nutrition supplements will be assessed at each clinic visit.

Biomarkers will be analyzed at randomization, and weeks 4 and 8 after randomization. Additionally, measurements of resource utilization will be measured such as the number of hospital days for non-chemotherapy-related problems, the number of sick visits to the clinic, dietitian visits, infections, and rates of relapse or overall survival. Biomarkers will be drawn when the children are in the clinic for chemotherapy or lab work. The participants will already have their central venous line accessed by a qualified clinic RN and labs will be drawn at that time to ensure no extra harm to the patient. Additionally, all patients will have EMLA cream used to numb the area prior to having a clinic RN who is trained in accessing ports and has accessed the ports during previous clinic visits and will continue to do so throughout therapy.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of pediatric cancer

Exclusion Criteria:

* Current use or history of enteral nutrition, oral supplement, or orexigenic/anorectic use.

Ages: 2 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 19 (Actual)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-08-04 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Body Composition | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  Change in body composition will be measured by ultrasound of the quadricep muscle layer thickness in millimeters.
Body Composition | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  Change in body composition will be measured by mid-upper arm circumference via z-scores by measuring the mid-upper arm in centimeters and comparing to CDC standards.

SECONDARY OUTCOMES:
Intolerances to interventions | Those randomized to a treatment group, will receive measurements at randomization and 1 & 3 months.
  These will be measured by CTCAEs to determine grade toxicity from interventions.
Change in weight | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  This will be measured with weight in kilograms and will be combined with data from CDC standardized growth charts to provide the weight z-score.
Change in BMI | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  This will be measured with pediatric z-scores for BMI and weight/length z-scores. Weight in kilograms and height in cm will be combined to report BMI in kg/m^2 and then plotted on CDC growth charts for z-scores.
Biomarkers | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These biomarkers will be measured via central venous lines, including IL-6 (pg/mL)
Biomarkers | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These biomarkers will be measured via central venous lines, including leptin (ng/mL) and vitamin D (ng/mL).
Biomarkers | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These biomarkers will be measured via central venous lines, including lipid profile (mg/dL).
Biomarkers | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These biomarkers will be measured via central venous lines, including cystatin-c (mg/L) and CRP (mg/L).
Physical Activity | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  Physical activity will be measured by team assessment of Lanksy Play-Performance Scale for Pediatric Functional Status. This scale uses parent descriptions of child's activity to assess ability and response to treatment. Scale ranges from 0-100 with a higher score indicating greater activity.
Tube feeding compliance | Those randomized will receive measurements at randomization and 1 & 3 months.
  Compliance will be analyzed by self-reported weekly compliance tube feeding volume which will be measured by the change in volume in mL compared to prescribed amounts in mL.
Oral nutrition supplements compliance | Those randomized will receive measurements at randomization and 1 & 3 months.
  Compliance will be analyzed by self-reported weekly compliance oral nutrition supplements which will be measured by the change in volume in number of cans compared to prescribed amounts in number of cans.
Medication compliance | Those randomized will receive measurements at randomization and 1 & 3 months.
  Compliance will be analyzed by self-reported weekly compliance of medication consumption which will be measured by the change in days all prescribed medications were taken compared to days where less medications than prescribed were taken.
Clinical measures | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These measurements will include the number of days hospitalized for nutrition-related issues
Clinical measures | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These measurements will include the number of clinic visits for nutrition-related issues
Clinical measures | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These measurements will include if they have a diagnosis of malnutrition (yes/no).
Clinical measures | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These measurements will include the rate of relapse or progression (yes/no)
Clinical measures | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These measurements will include the number of days that cancer treatment is put on hold.
Clinical measures | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These measurements will include the presence of chemotherapy toxicities using CTCAE (Common Terminology Criteria for Adverse Events) grading scale (grades 1-4)
Clinical measures | Baseline, at 3 and 6 months from baseline for control group. Those randomized will receive measurements at randomization and 1 & 3 months.
  These measurements will include the diagnosis type (cancer type).

CONTACTS AND LOCATIONS:
Overall Officials: Corey J Hawes, DCN, RD, CSO, CNSC, LD, Principal Investigator — University of Kentucky, Kentucky Children's Hospital
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/73/NCT06175273/ICF_000.pdf